CLINICAL TRIAL: NCT01837368
Title: Research Project About Psychological Strain, Quality of Life and Emotional Awareness in Patients With Tinnitus
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: tinnitus_T0
Record Dates: First submitted 2012-12-19; First posted 2013-04-23 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational research — It is a observational research, no intervention are performed

SUMMARY:
Validation of PRISM (Pictorial Representation of Illness and Self Measure) as a assessment of quality of life and suffering in patients with tinnitus.

Association between experiencing, verbalizing and regulating emotions and perceived tinnitus.

Correlation analysis are used to search for connections between the subjective behavioral outcomes mentioned above and the objective EEG-patterns.

DETAILED DESCRIPTION:
Validation of PRISM (Pictorial Representation of Illness and Self Measure). Assessment of quality of life and suffering in patients with tinnitus in an observational study using different questionnaires. (THI, TF, TBF-12, BDI, BAI, SF-36).

THI - Tinnitus Handicap Inventory

TF - Tinnitus Questionnaire after Goebel and Hiller

TBF-12 - Tinnitus Impairment Questionnaire

BDI - Beck Depression Inventory

BAI - Beck Anxiety Inventory

SF-36 - Short Form 36 Health Survey Questionnaire

Association between experiencing, verbalizing and regulating emotions and perceived tinnitus using the TAS-20 (20-Item Toronto Alexithymia Scale) and the above mentioned questionnaires.

EEG-studies on the spontaneous brain activity of individuals affected by tinnitus consistently report differences in the composition of the EEG-frequency spectrum between individuals with tinnitus and healthy controls. Furthermore it has been shown that not only the auditory cortex but other regions of the brain are involved in the perception of the chronic ear noise as well. Among them is the limbic system which is associated with the emotional processing of the human brain.

Correlation analysis are used to search for connections between the subjective behavioral outcomes mentioned above and the objective EEG-patterns. Aim of the current study is to provide conclusive models of associated assessments of the psychological strain end emotional stress of individuals suffering from tinnitus and objective EEG-analysis.

ELIGIBILITY:
Inclusion criteria:

* all patients older than 18 years with tinnitus who want to participate the investigation during the period of data acquisition

Exclusion criteria:

* patients younger than 18 years,
* insufficient knowledge of the German language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tinnitus
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Values of PRISM | 4 weeks
  measures the burden of suffering
TAS | 4 weeks
  Alexithymia- measured with TAS-toronto alexithymia scale; measures ability to identify feelings, describe feeling, and style of thinking

SECONDARY OUTCOMES:
Quality of life (SF-36), perceived grade of tinnitus (THI, TF, TBF-12) and the clinical characteristic of tinnitus. | 4 weeks
  composite outcome
comorbidities | 4 weeks
  measured with BAI , BDI
Tinnitus functional index (TFI) perceived grade of tinnitus | 4 weeks
  Composite outcome

CONTACTS AND LOCATIONS:
Overall Officials: Steffi Weidt, MD, Principal Investigator — University Hospital Zurich, Division of Psychiatry and Psychotherapy
Locations (1):
- University Hospital Zurich, Division of Psychiatry and Psychotherapy, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Peter N, Kleinjung T, Jeker R, Meyer M, Klaghofer R, Weidt S. Tinnitus functional index: validation of the German version for Switzerland. Health Qual Life Outcomes. 2017 May 5;15(1):94. doi: 10.1186/s12955-017-0669-x. PMID 28476163
- See also: Publication Tinnitus and PRISM — http://www.ncbi.nlm.nih.gov/pubmed/?term=PRISM+Tinnitus
- See also: Publication Tinnitus and quality of life — http://www.ncbi.nlm.nih.gov/pubmed/26850646